CLINICAL TRIAL: NCT00686010
Title: A 4-Weeks Treatment, Randomised, Double-Blind, Parallel-Group Study Evaluating The Efficacy and Safety of JTT-705 300 to 900mg in Comparison With Placebo in Patients With Type II Hyperlipidaemia
Brief Title: Efficacy and Safety of JTT-705 300, 600 And 900mg in Comparison With Placebo in Patients With Type II Hyperlipidaemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Japan Tobacco Inc. (Industry)
Responsible Party: Yukio N, Clinical Research Planning Dept., General Manager, Japan Tobacco Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAY2-1
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Type II Hyperlipidaemia
Keywords: CETP Inhibitor; HDL-C; LDL-C; Apolipoprotein
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — dalcetrapib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): JTT-705 300mg
  Interventions: Drug: JTT-705 300mg
- 3 (Experimental): JTT-705 600mg
  Interventions: Drug: JTT-705 600mg
- 4 (Experimental): JTT-705 900mg
  Interventions: Drug: JTT-705 900mg

INTERVENTIONS:
Drug: Placebo — Placebo tablet, 3 tablets, oral, once daily after breakfast
  Arms: 1
Drug: JTT-705 300mg — JTT-705 tablet, 1 tablet, oral, once daily, after breakfast. Placebo tablet, 2 tablets, oral, once daily, after breakfast.
  Arms: 2
Drug: JTT-705 600mg — JTT-705 tablet, 2 tablets, oral, once daily, after breakfast. Placebo tablet, 1 tablet, oral, once daily, after breakfast
  Arms: 3
Drug: JTT-705 900mg — JTT-705 tablet, 3 tablets, oral, once daily, after breakfast
  Arms: 4

SUMMARY:
To demonstrate the effect of JTT-705 doses from 300 mg to 900 mg on the elevation of HDL-C and on the inhibition of CETP activity versus placebo, in patients presenting with mild dyslipidaemia. These objectives will be tested after 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with of Type II hyperlipidaemia
* Patients having lipid values as indicated below:

  * HDL-C < 1.6 mmol/l
  * TG < 4.5 mmol/l
* Male and females between 18 and 65 years old (If female must be post-menopausal, or pre-menopausal and surgically sterile or using an acceptable form of contraception)

Exclusion Criteria:

* Body Mass Index (BMI) > 35 kg/m²
* Pregnant, breast feeding, or woman with child bearing potential without an effective method of contraception
* Concomitant use of medications identified in the protocol

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2000-05; Primary Completion 2001-01 (Actual); Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
%change from baseline in HDL-C, Inhibition of CETP activity | 4-weeks

SECONDARY OUTCOMES:
%change from baseline in LDL-C and TC/HDL ratio | 4-weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam, Utrecht, Rotterdam, Nijmegen, Arnhem, Groningen, Dordrecht, Hoorn, Groningen, Amsterdam, Netherlands